CLINICAL TRIAL: NCT04706741
Title: A Phase 2 Trial of the Efficacy and Safety of the Interleukin-17A Inhibitor Izokibep (ABY-035) in the Treatment of Non-infectious Intermediate, Posterior or Pan-uveitis (LINNAEA)
Brief Title: A Trial of the Efficacy and Safety of Izokibep in the Treatment of Non-anterior Uveitis
Acronym: LINNAEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABY-035-203
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-08

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Prednisone; Prednisolone

STUDY DESIGN:
Intervention Model Description: The primary purpose of the study is treatment of active Noninfectious Intermediate, Posterior or Pan-uveitis
  The study includes one treatment arm, into which 10 patients are planned to be enrolled
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Izokibep and maintenance corticosteroid dose (Experimental): Izokibep+ Prednisolon/Prednisone
  Interventions: Drug: Izokibep; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Izokibep — Izokibep is an Interleukin-17 Inhibitor that will be administered subcutaneously
  Other Names: ABY-035
Drug: Prednisone/Prednisolone — Background Corticosteroid
  Other Names: Prednisone

SUMMARY:
This is a multicenter, phase 2 trial to explore the efficacy and safety of Izokibep (ABY-035) in treating disease activity in patients with non-Infectious Intermediate, Posterior, Pan-Uveitis with significant disease activity at BL despite treatment with stable doses of corticosteroids (≥7 to ≤40 mg/day oral prednisolon or equivalent).

DETAILED DESCRIPTION:
This is a multicenter, phase 2 trial to explore the efficacy and safety of Izokibep (ABY-035) in treating disease activity in patients with non-Infectious Intermediate, Posterior, Pan-Uveitis with significant disease activity at BL despite treatment with stable doses of corticosteroids (≥7 to ≤40 mg/day oral prednisolon or equivalent).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at SCR
2. Previously documented medical history with diagnosed unilateral or bilateral NIIPPU
3. Active disease at BL defined by the presence of at least 1 of the following criteria in at least one eye despite treatment with stable doses of corticosteroids for at least 2 weeks:

   1. Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion by Dilated Indirect Ophthalmoscopy (DIO), Fundus Photography, Fluorescein angiography (FA), spectral-domain optical coherence tomography (SD-OCT) to determine whether a lesion is active or inactive (the central reader's assessment using FA, FP, and or SD-OCT is required to confirm eligibility).
   2. ≥2+ vitreous haze ( NEI/SUN criteria) by DIO and Fundus Photography (the central reader's assessment using Fundus Photography is required to confirm eligibility).
4. On treatment with oral corticosteroids (≥7 to ≤40 mg/day oral prednisolon or equivalent) at a stable dose for at least 2 weeks before BL

Exclusion Criteria:

1. Subject with isolated anterior uveitis
2. Subject with Occlusive Behçet's disease, Acute Posterior Multifocal Placoid Pigment Epitheliopathy, Acute Posterior Pigment Epithelitis, Multiple Evanescent White Dot Syndrome, Punctate Inner Choroiditis or serpiginous choroidopathy
3. Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, syphilis, cytomegalovirus, Lyme disease, toxoplasmosis, Human T-Lymphotropic Virus Type 1 infection, Whipple's disease, herpes zoster virus, and herpes simplex virus
4. Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial
5. Planned (elective) eye surgery within 80 weeks after BL
6. History of prior refractive laser surgery, retinal laser photocoagulation, or neodymium-doped yttrium aluminium garnet posterior capsulotomy within 30 days before BL
7. History of any other prior ocular surgery within 90 days before BL
8. Subject with intraocular pressure (IOP) of ≥25 mmHg while on ≥2 glaucoma medications or evidence of glaucomatous optic nerve injury
9. Subject with severe vitreous haze that precludes visualization of the fundus at BL
10. Subject has a contraindication for mydriatic eye drops OR subject cannot be dilatated sufficiently well to permit good fundus visualization
11. Subject with BCVA <20 letters (ETDRS) in at least one eye at BL
12. Subject with intermediate uveitis or panuveitis who has presence or history of whitish exudates on the inferior pars plana (snowbanking) or vitreal inflammatory aggregates (snowballs) in combination with a medical history or signs or symptoms suggestive of a demyelinating disease such as multiple sclerosis
13. Subject with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy
14. Subject with neovascular/wet age-related macular degeneration
15. Subject with an abnormality of the vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process
16. Subject with a history of active scleritis within 12 months of SCR Criteria that relate to comorbidity
17. Uncontrolled inflammatory bowel disease
18. Infection requiring treatment with IV anti-infectives within 30 days before BL or oral anti-infectives within 14 days before BL
19. Subject with any active infection that based on the investigator's clinical assessment makes the subject an unsuitable candidate for the trial
20. History or any signs of lymphoproliferative disease, or a known malignancy or a history of malignancy within the previous 3 years (except for basal cell or squamous cell carcinoma of the skin that had been fully excised with no evidence of recurrence) Criteria that relate to laboratory testing
21. A positive test for subclinical/latent TB infection (i.e. positive QuantiFERON®-TB Gold test or equivalent product) suggestive of TB at SCR will require that the subject is thoroughly evaluated for active tuberculosis. If the subject is diagnosed with latent TB and active TB can be ruled out, the subject can be included if the subject has gone through an adequate course of prophylaxis as per local standard of care 12 weeks prior to SCR.
22. Positive Fluorescent treponemal (FTA)- absorption test (syphilis)
23. Subject with intolerance to high-dose oral corticosteroids (equivalent to oral prednisolon 1 mg/kg/day or 60 mg/day)
24. The subject has received any biologic therapy (including ABY-035 or any other IL-17i or IL-17 receptor inhibitor, e.g. secukinumab, ixekizumab, brodalumab or anti-TNF-alpha therapy) within 8 weeks before BL.
25. Subject on >1 concomitant non-biologic NCSIT
26. Subject on 1 concomitant non-biologic NCSIT:

    a) But the medication is not listed as permissible b) The medication is listed as permissible, but the dose has not been stable within the last 3 months before BL c) The medication is listed as permissible, but the dose exceeds the allowable level; to be acceptable, the dose needs to be: i) Methotrexate (MTX) ≤25 mg/week ii) CsA ≤4 mg/kg/day iii) Mycophenolate mofetil ≤2 grams/day or an equivalent drug to mycophenolate mofetil (e.g., mycophenolic acid) at an equivalent dose approved by the Medical monitor iv) Azathioprine ≤175 mg/day v) Tacrolimus (oral formulation) ≤8 mg/day

28] The subject has received Retisert®, Iluvien®, or Yutiq® (glucocorticosteroids implant) within 3 years before BL or who has had complications related to the device. The subject has had any of these glucocorticosteroids implant (glucocorticosteroid implant) removed within 90 days before BL or has had complications related to the removal of the device 29] The subject has received intraocular or periocular corticosteroids within 90 days before BL 30] The subject has received Ozurdex® (dexamethasone implant) within 6 months before BL 31] The subject has received intravitreal methotrexate within 90 days before BL 32] The subject has received intravitreal anti- Vascular Endothelial Growth Factor (VEGF) therapy:

1. within 45 days of BL for Lucentis® (ranibizumab) or Avastin® (bevacizumab)
2. or within 60 days of BL for anti-VEGF Trap (aflibercept)
3. or within 84 days of BL for Beovu® (brolucizumab) 33] Subject on systemic carbonic anhydrase inhibitor within 1 week before SCR 34] Subject on cyclophosphamide within 30 days before BL 35] Prior or current use of chlorambucil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Complete Response | BL to Week 10
  Complete Response is defined as Yes/No by visit by meeting at least 1 of the following criteria in at least one eye:
  1. Inflammatory, chorioretinal and/or inflammatory retinal vascular lesions - No such active lesions; all prior lesions appear inactive
  2. ACC Count - Trace or absent (0.5+ or 0)
  3. Vitreous Haze - Trace or absent (0.5+ or 0)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Betah, MD, Study Director — ACELYRIN Inc.
Locations (4):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Hagerstown, Maryland
  - Research Site, Plano, Texas